CLINICAL TRIAL: NCT05831943
Title: Low Tube Voltage Kidney Computed Tomography Using Low Concentration Iodine Contrast Agent: A Comparison Study With Conventional CT Protocol
Brief Title: A Study on the Verification of Kidney CT Non-inferiority Using Low Concentration Contrast Agent
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Taejoon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, June Young Seo, Clinical fellow, Seoul National University Hospital
Other Study IDs: SNUH-2022-0218
Record Dates: First submitted 2023-04-16; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Renal Disease
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Renal CT evaluation: Patients who are planned kidney contrast enhanced CT scan
  Interventions: Diagnostic Test: Contrast enhanced Kidney CT

INTERVENTIONS:
Diagnostic Test: Contrast enhanced Kidney CT — * Test group : Patient undergoing CT scan with 80kVP protocol and using low concentration intravascular contrast media ( Iobrix 270 mgl/MI , Taejoon pharm, Seoul, South Korea)
  * Control group : Patient undergoing CT scan with 120kVP protocol and using high concentration intravascular contrast media ( Iobrix 320 mgl/MI , Taejoon pharm, Seoul, South Korea)

SUMMARY:
This prospective study aims to evaluate clinical usefulness of low-voltage renal CT using low-concentration contrast agent and to compare with existing imaging techniques.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with no abnormalities in renal function (Serum creatinine < 1.4 mg/dl , GFR > 45mL/min/1.73 m2) in blood tests performed within one month
* Those who understand the contents of the research subject explanation and voluntarily sign the consent form

Exclusion Criteria:

* Body mass index > 30
* Subjects whose renal function abnormality was confirmed in a blood test (Serum creatinine > 1.4 mg/dl , GFR < 45mL/min/1.73 m2) conducted within one month
* Diabetic patients taking metformin
* Those with a history of urinary tract obstruction
* Those with a history of bladder, urinary tract, or kidney surgery that may affect the evaluation of the contrast agent in the renal parenchyma
* Those whose anatomical deformities have been identified in previous images that may interfere with image analysis
* Those who know or have been reported to have a history of contrast agent side effects in previous CT scans
* Those with a history of hypersensitivity or adverse reactions to iobrix (intravascular CT contrast) or iodine based agent
* Those with severe thyroid disease
* Pregnancy
* Those who are judged unsuitable for clinical trials by the researcher for reasons such as having other severe diseases or being judged to have a high risk of adverse reactions to intravascular contrast agents

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who need contrast enhanced CT scan for anatomical evaluation of kidney
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Quantitative analysis - Radiation dose | 6 months after the CT scan
  Effective radiation dose (mSv) annotated on CT image
Quantitative analysis - Signal to noise ratio | 6 months after the CT scan
  Value calculated by ( mean attenuation / standard deviation of attenuation of contrast area)
Quantitative analysis - Contrast to noise ratio | 6 months after the CT scan
  Value calculated by [ ( mean attenuation - attenuation of contrast area) / standard deviation of attenuation of contrast area ]
Qualitative analysis - Diagnostic acceptability, Noise , Artifacts , Sharpness | 6 months after the CT scan
  4 points scale quantitative analysis evaluated by three different radiologists

SECONDARY OUTCOMES:
Diagnoses of focal lesion and inter-observer agreement | 6 months after the CT scan
  Detection by three individual radiologist and its inter-observer agreement

CONTACTS AND LOCATIONS:
Overall Officials: June Young Seo, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Jong-no Gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choi MH, Lee YJ, Jung SE. The Image Quality and Diagnostic Performance of CT with Low-Concentration Iodine Contrast (240 mg Iodine/mL) for the Abdominal Organs. Diagnostics (Basel). 2022 Mar 19;12(3):752. doi: 10.3390/diagnostics12030752. PMID 35328304
- [Background] Yoo YJ, Choi IY, Yeom SK, Cha SH, Jung Y, Han HJ, Shim E. Evaluation of Abdominal CT Obtained Using a Deep Learning-Based Image Reconstruction Engine Compared with CT Using Adaptive Statistical Iterative Reconstruction. J Belg Soc Radiol. 2022 Apr 8;106(1):15. doi: 10.5334/jbsr.2638. eCollection 2022. PMID 35480337
- [Background] Ichikawa S, Motosugi U, Shimizu T, Kromrey ML, Aikawa Y, Tamada D, Onishi H. Diagnostic performance and image quality of low-tube voltage and low-contrast medium dose protocol with hybrid iterative reconstruction for hepatic dynamic CT. Br J Radiol. 2021 Dec;94(1128):20210601. doi: 10.1259/bjr.20210601. Epub 2021 Sep 29. PMID 34586900
- [Background] Kim SY, Cho JY, Lee J, Hwang SI, Moon MH, Lee EJ, Hong SS, Kim CK, Kim KA, Park SB, Sung DJ, Kim Y, Kim YM, Jung SI, Rha SE, Kim DW, Lee H, Shim Y, Hwang I, Woo S, Choi HJ. Low-Tube-Voltage CT Urography Using Low-Concentration-Iodine Contrast Media and Iterative Reconstruction: A Multi-Institutional Randomized Controlled Trial for Comparison with Conventional CT Urography. Korean J Radiol. 2018 Nov-Dec;19(6):1119-1129. doi: 10.3348/kjr.2018.19.6.1119. Epub 2018 Oct 18. PMID 30386143
- [Background] Taguchi N, Oda S, Utsunomiya D, Funama Y, Nakaura T, Imuta M, Yamamura S, Yuki H, Kidoh M, Hirata K, Namimoto T, Hatemura M, Kai N, Yamashita Y. Using 80 kVp on a 320-row scanner for hepatic multiphasic CT reduces the contrast dose by 50 % in patients at risk for contrast-induced nephropathy. Eur Radiol. 2017 Feb;27(2):812-820. doi: 10.1007/s00330-016-4435-y. Epub 2016 May 30. PMID 27240454
- [Background] Zhang H, Ma Y, Lyu J, Yang Y, Yuan W, Song Z. Low kV and Low Concentration Contrast Agent with Iterative Reconstruction of Computed Tomography (CT) Coronary Angiography: A Preliminary Study. Med Sci Monit. 2017 Oct 20;23:5005-5010. doi: 10.12659/msm.904251. PMID 29051477
- [Background] Botsikas D, Barnaure I, Terraz S, Becker CD, Kalovidouri A, Montet X. Value of liver computed tomography with iodixanol 270, 80 kVp and iterative reconstruction. World J Radiol. 2016 Jul 28;8(7):693-9. doi: 10.4329/wjr.v8.i7.693. PMID 27551339
- [Background] Park IK, Park J, Kim TH, Lee J, Han K, Oh C, Park CH. Non-inferior low-dose coronary computed tomography angiography image quality with knowledge-based iterative model reconstruction for overweight patients. PLoS One. 2018 Dec 26;13(12):e0209243. doi: 10.1371/journal.pone.0209243. eCollection 2018. PMID 30586449
- [Background] Hwang I, Cho JY, Kim SY, Oh SJ, Ku JH, Lee J, Kim SH. Low tube voltage computed tomography urography using low-concentration contrast media: Comparison of image quality in conventional computed tomography urography. Eur J Radiol. 2015 Dec;84(12):2454-63. doi: 10.1016/j.ejrad.2015.09.010. Epub 2015 Sep 10. PMID 26388465
- [Background] Mayer C, Meyer M, Fink C, Schmidt B, Sedlmair M, Schoenberg SO, Henzler T. Potential for radiation dose savings in abdominal and chest CT using automatic tube voltage selection in combination with automatic tube current modulation. AJR Am J Roentgenol. 2014 Aug;203(2):292-9. doi: 10.2214/AJR.13.11628. PMID 25055262
- [Background] Araki K, Yoshizako T, Yoshida R, Tada K, Kitagaki H. Low-voltage (80-kVp) abdominopelvic computed tomography allows 60% contrast dose reduction in patients at risk of contrast-induced nephropathy. Clin Imaging. 2018 Sep-Oct;51:352-355. doi: 10.1016/j.clinimag.2018.05.027. Epub 2018 Jun 9. PMID 29982133